CLINICAL TRIAL: NCT03272035
Title: General Practitioners' Felt With Their Patients' Death (REGIDAQ)
Acronym: REGIDAQ
Status: Completed | Type: Observational
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: I16018 (REGIDAQ)
Record Dates: First submitted 2017-08-23; First posted 2017-09-05 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2017-08

CONDITIONS: Death
Keywords: General practice; death; bereavement
MeSH Terms: conditions — Death

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Very few studies are dealing with the way general practitioners feel the death of their patients. Main studies about that subject are qualitative. It needs quantitative studies to analyse how is felt general practitioners' patients' death. This is an epidemiologic quantitative cross-sectional study. The Studied population is the whole of the general practitioners of the region Nouvelle-Aquitaine. The primary endpoint is the percentage of the general practitioners which have hard time living with their patients' death. The secondary endpoints are to evaluate the general practitioners' help needing after their patients' death, to evaluate the personal and professional impact of the patient's death, the percentage of general practitioners using chemical aid after their patients' death and to determinate the existence of support facilities to help general practitioners to stand patients' death. The results of that study could help general practitioners to improve their medical practice in the patient's death situation.

ELIGIBILITY:
Inclusion Criteria:

* General practitioners from the Nouvelle-Aquitaine region.
* Exclusive or joint exercise of general medicine.
* None retired

Exclusion Criteria:

* Retired patricians
* Students, Residents
* General practitioners from another region
* General practitioners with no general medicine activity

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: General practitioners from the Nouvelle Aquitaine region
Sampling Method: Non-Probability Sample
Enrollment: 481 (Actual)
Dates: Start 2018-02-13 (Actual); Primary Completion 2018-05-13 (Actual); Study Completion 2018-05-13 (Actual)

PRIMARY OUTCOMES:
percentage of hard time living | 2 months (End of study)
  percentage of general practitioners which have hard time living with their patients' death

SECONDARY OUTCOMES:
percentage of help needing | 2 months (End of study)
  percentage of general practitioners which need help after their patients' death
percentage of personal impact | 2 months (End of study)
  percentage of general practitioners which have a personal impact when their patient's death
percentage of professional impact | 2 months (End of study)
  percentage of general practitioners witch have a professional impact when the patient's death
percentage of chemical aid using | 2 months (End of study)
  percentage of general practitioners using chemical aid after their patients' death
support facilities | 2 months (End of study)
  Determinate the existence of support facilities to help general practitioners to stand patients' death

CONTACTS AND LOCATIONS:
Overall Officials: Karen Rudelle, doctor, Principal Investigator — University Hospital, Limoges
Locations (1):
- University Hospital, Limoges, France